CLINICAL TRIAL: NCT06405048
Title: Evaluating the Feasibility and Effectiveness of a Mock-up Fact-checking Extension to Improve Ability to Debunk HPV Vaccine Misinformation Among Parents of Middle School Girls: A Survey Experiment
Brief Title: Impact of a Mock-up Fact-checking Extension on HPV Vaccine Misinformation: A Survey Experiment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zhiyuan Hou, Associate Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Fact-checking Extension
Record Dates: First submitted 2024-04-26; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: HPV Vaccine
Keywords: HPV vaccine; knowledge; misinformation; vaccine confidence; fact-checking extension
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mock-up fact-checking extension intervention group (Experimental): Intervention group participants will engage with three modules:
  In Module 1, participants will examine six Weibo post screenshots, each featuring a mock-up of a Chinese fact-checking extension. Participants in the intervention group will assess a statement linked to the content of each post, which aligns with predefined HPV vaccine knowledge from section (b). Their response options will be: 1) Correct, 2) Incorrect, or 3) I don't know, taking into account both the post and the extension's feedback.
  In the module 2, participants will review four additional Weibo post screenshots, two of which include false information. Responses will follow the same format used in Module 1.
  In Module 3, participants will choose whether to view Weibo post screenshots with the fact-checking extension enabled or disabled. If they choose "Yes", the screenshot will be displayed with the extension; if "No", it will be shown without the extension.
  Interventions: Other: Mobile Weibo post screenshot with mock-up Chinese fact-checking extension
- Control group (No Intervention): Control group participants will participate in three modules:
  In Modules 1 and 2, they will review six and four Weibo post screenshots, respectively, without the mock-up Chinese fact-checking extension. Participants will evaluate statements linked to the content of each post, aligning with predefined HPV vaccine knowledge from section (b). Their response options will be: 1) Correct, 2) Incorrect, or 3) I don't know, based solely on the content of the posts.
  In Module 3, participants will choose whether to view Weibo post screenshots with the fact-checking extension enabled or disabled. If they choose "Yes", the screenshot will be displayed with the extension; if "No", it will be shown without the extension.

INTERVENTIONS:
Other: Mobile Weibo post screenshot with mock-up Chinese fact-checking extension — The intervention in this survey experiment involves mobile Weibo post screenshots equipped with a mock-up Chinese fact-checking browser extension. All screenshots are based on actual Weibo posts. The fact-checking content is generated by a Large Language Model (LLM), tailored to relevant knowledge and prompts, and subsequently validated by experts. The Weibo posts cover a range of popular topics known to contain misinformation, including infertility, safety, vaccine ingredients, high-risk cervical cancer types, regular check-ups, transmission routes, and others.
  Arms: Mock-up fact-checking extension intervention group

SUMMARY:
The primary objective of this survey experiment study is to measure the impact of a mock-up Chinese fact-checking extension on the ability to dispel HPV and HPV vaccine-related misinformation among parents of middle school girls in China.

DETAILED DESCRIPTION:
This survey experiment study aims to assess the feasibility and effectiveness of a mock-up Chinese fact-checking extension on improving the ability to identify HPV and HPV vaccine-related misinformation among parents of middle school girls in three economically diverse regions of China. This includes Shanghai megacity, an urban city in Anhui Province, and rural counties in Anhui Province. The participants will be parents of middle school girls who have not yet received the HPV vaccine. This experiment will randomly assign the participants into intervention or control group. Participants in the intervention group will use a mock-up Chinese fact-checking extension whereas those in control group will not.

The sample size for this study was determined based on the two primary outcomes: knowledge of the HPV vaccine and the ability to dispel misinformation. A review of the existing literature suggests that the intention or confidence among Chinese parents to vaccinate their children with the HPV vaccine, as well as their knowledge about the vaccine and capability to counteract misinformation, typically ranges from 50% to 70%. We assumed a baseline rate of 60% for both vaccine knowledge and misinformation discernment. It is anticipated that exposure to educational interventions will increase these rates by 10%, elevating them to 70%. Using a significance level of 0.05 and a statistical power of 90%, the required sample size was calculated to be a minimum of 473 participants per group. To accommodate potential variability and to strengthen the robustness of the study, 500 participants will be recruited for each group, maintaining a 1:1 ratio. This approach results in a total sample size of 1,000 participants. Such a sample size ensures that the study is sufficiently powered to detect a significant change in the outcomes of interest.

In this study, 11 mobile Weibo post screenshots were created, covering a range of topics including infertility, safety, vaccine ingredients, high-risk cervical cancer types, regular check-ups, transmission routes, and others.

The participants in both groups will complete a questionnaire consisting of six phases:

1. Phase 1 (Baseline Assessment): Participants in both the intervention and control groups will complete a questionnaire covering (a) basic demographic information, (b) HPV vaccine knowledge, (c) HPV vaccine awareness and confidence, and (d) vaccination intentions.
2. Phase 2 (Intervention Module 1): Participants in the intervention group will review six Weibo post screenshots, each featuring a mock-up Chinese fact-checking extension. The control group will view identical screenshots, but without the fact-checking extension. Half of these posts will include false information. After viewing each post, those in the intervention group will evaluate a statement related to the Weibo content and corresponding to one of the predefined (b) HPV vaccine knowledge. Their responses will be: 1) Correct, 2) Incorrect, or 3) I don't know, considering both the post content and the fact-checking extension's findings. Participants in the control group will assess the same statement based only on the post content, with the same response options.
3. Phase 3 (Intervention Module 2): All participants will review four additional Weibo post screenshots, including two containing false information, to evaluate whether exposure to the mock-up fact-checking extension has improved the intervention group's ability to identify false information. The same question format from Intervention Module 1 will be used for responses.
4. Phase 4 (Post-intervention Assessment): All participants are required to fill out sections on (c) HPV vaccine awareness and confidence, and (d) vaccine intentions.
5. Phase 5 (Intervention Module 3): All participants in both groups will be asked whether they use a mock-up fact-checking extension when viewing Weibo post screenshots. If participants choose 'Yes', they will view a Weibo post screenshot with the extension displayed; if they choose 'No', the extension will not be displayed. The same question format from Intervention Module 1 will be used for responses. This phase aims to assess participants' behaviour regarding the use of the extension.
6. Phase 6 (User Experience Assessment): All participants will complete the section (e) the user experience with a mock-up fact-checking extension.

Following the completion of the experiment, a debunking procedure will be conducted for participants in both the intervention and control groups. This is to avoid any potential risks associated with the spread of misinformation on Weibo.

Data analysis will employ Difference-in-Differences (DID) analysis, multiple logistic regression, and other suitable statistical methods to evaluate the effectiveness of the mock-up Chinese fact-checking extension.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be parents or legal guardians of female students currently enrolled in participating middle school.
2. The parent's or guardian's female middle school student must not have received the HPV vaccine, must not have an HPV vaccination appointment scheduled, and must not have any contraindications to receiving the HPV vaccine.
3. Participants must be free of mental health disorders or visual/reading disabilities that could prevent their full participation in and completion of the intervention activities.
4. Participants must have provided informed consent and expressed a willingness to actively participate throughout the study.

Exclusion criteria are defined as individuals not meeting the aforementioned inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-28 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Ability to debunk misinformation | Day 1, in a single survey
  This outcome measures participants' ability to debunk misinformation about the HPV or HPV vaccine. Total debunking scores range from 0 to 10, with higher scores reflecting better debunking skills.

SECONDARY OUTCOMES:
HPV vaccination intention | Day 1, in a single survey
  Intention to vaccinate daughters against HPV, measured on a five-point Likert scale from 0 ("very unwilling") to 5 ("very willing").
HPV vaccine confidence | Day 1, in a single survey
  Vaccine Confidence Index (VCI), including confidence on vaccine effectiveness and safety, measured on a five-point Likert scale from 0 ("strongly disagree") to 5 ("strongly agree").
Tool acceptance | Day 1, in a single survey
  Determines whether participants would like to use a mock-up fact-checking extension when viewing screenshots of Weibo posts. Responses are either Yes (1) or No (0).
User experience of mock-up fact-checking extension | Day 1, in a single survey
  4 questions about the user experience of a mock-up fact-checking browser extension, measured using a five-point Likert scale from "strongly disagree" to "strongly agree"

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyuan Hou, PhD, Principal Investigator — Fudan University; Leesa Lin, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- China (2):
  - Chizhou Health Center for Disease Control and Prevention, Chizhou, Anhui
  - Jiading District Center for Disease Control and Prevention, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices), will be shared upon reasonable requests. A written data-sharing request for meta-analysis should be submitted by email with a methodologically sound proposal. Proposals should be directed to zyhou@fudan.edu.cn; to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal for meta analysis. Proposals should be directed to zyhou@fudan.edu.cn; to gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Lee KY, Dabak SV, Kong VH, Park M, Kwok SLL, Silzle M, Rachatan C, Cook A, Passanante A, Pertwee E, Wu Z, Elkin JA, Larson HJ, Lau EHY, Leung K, Wu JT, Lin L. Effectiveness of chatbots on COVID vaccine confidence and acceptance in Thailand, Hong Kong, and Singapore. NPJ Digit Med. 2023 May 25;6(1):96. doi: 10.1038/s41746-023-00843-6. PMID 37231110
- [Background] Huang S, Yang J, Fong S, Zhao Q. Artificial intelligence in the diagnosis of COVID-19: challenges and perspectives. Int J Biol Sci. 2021 Apr 10;17(6):1581-1587. doi: 10.7150/ijbs.58855. eCollection 2021. PMID 33907522
- [Background] Scherer LD, McPhetres J, Pennycook G, Kempe A, Allen LA, Knoepke CE, Tate CE, Matlock DD. Who is susceptible to online health misinformation? A test of four psychosocial hypotheses. Health Psychol. 2021 Apr;40(4):274-284. doi: 10.1037/hea0000978. Epub 2021 Mar 1. PMID 33646806
- [Background] Bin Naeem S, Kamel Boulos MN. COVID-19 Misinformation Online and Health Literacy: A Brief Overview. Int J Environ Res Public Health. 2021 Jul 30;18(15):8091. doi: 10.3390/ijerph18158091. PMID 34360384
- [Background] Southwick L, Guntuku SC, Klinger EV, Seltzer E, McCalpin HJ, Merchant RM. Characterizing COVID-19 Content Posted to TikTok: Public Sentiment and Response During the First Phase of the COVID-19 Pandemic. J Adolesc Health. 2021 Aug;69(2):234-241. doi: 10.1016/j.jadohealth.2021.05.010. Epub 2021 Jun 22. PMID 34167883
- [Background] Tangcharoensathien V, Calleja N, Nguyen T, Purnat T, D'Agostino M, Garcia-Saiso S, Landry M, Rashidian A, Hamilton C, AbdAllah A, Ghiga I, Hill A, Hougendobler D, van Andel J, Nunn M, Brooks I, Sacco PL, De Domenico M, Mai P, Gruzd A, Alaphilippe A, Briand S. Framework for Managing the COVID-19 Infodemic: Methods and Results of an Online, Crowdsourced WHO Technical Consultation. J Med Internet Res. 2020 Jun 26;22(6):e19659. doi: 10.2196/19659. PMID 32558655
- [Background] Norman CD, Skinner HA. eHealth Literacy: Essential Skills for Consumer Health in a Networked World. J Med Internet Res. 2006 Jun 16;8(2):e9. doi: 10.2196/jmir.8.2.e9. PMID 16867972
- [Background] Hu D, Martin C, Dredze M, Broniatowski DA. Chinese social media suggest decreased vaccine acceptance in China: An observational study on Weibo following the 2018 Changchun Changsheng vaccine incident. Vaccine. 2020 Mar 17;38(13):2764-2770. doi: 10.1016/j.vaccine.2020.02.027. Epub 2020 Feb 22. PMID 32093982
- [Background] Chen L, Wang X, Peng TQ. Nature and Diffusion of Gynecologic Cancer-Related Misinformation on Social Media: Analysis of Tweets. J Med Internet Res. 2018 Oct 16;20(10):e11515. doi: 10.2196/11515. PMID 30327289
- [Background] Keelan J, Pavri V, Balakrishnan R, Wilson K. An analysis of the Human Papilloma Virus vaccine debate on MySpace blogs. Vaccine. 2010 Feb 10;28(6):1535-40. doi: 10.1016/j.vaccine.2009.11.060. Epub 2009 Dec 8. PMID 20003922
- [Background] Zimet GD, Rosberger Z, Fisher WA, Perez S, Stupiansky NW. Beliefs, behaviors and HPV vaccine: correcting the myths and the misinformation. Prev Med. 2013 Nov;57(5):414-8. doi: 10.1016/j.ypmed.2013.05.013. Epub 2013 May 31. PMID 23732252
- [Background] Huang Y, Xu S, Xu Y, Yao D, Wang L, Zhao Y, Wu Q. A New Strategy for Cervical Cancer Prevention Among Chinese Women: How Much Do They Know and How Do They React Toward the HPV Immunization? J Cancer Educ. 2021 Apr;36(2):386-394. doi: 10.1007/s13187-019-01642-y. PMID 31902089
- [Background] Zhang Y, Wang Y, Liu L, Fan Y, Liu Z, Wang Y, Nie S. Awareness and knowledge about human papillomavirus vaccination and its acceptance in China: a meta-analysis of 58 observational studies. BMC Public Health. 2016 Mar 3;16:216. doi: 10.1186/s12889-016-2873-8. PMID 26936076
- [Background] Li K, Li Q, Song L, Wang D, Yin R. The distribution and prevalence of human papillomavirus in women in mainland China. Cancer. 2019 Apr 1;125(7):1030-1037. doi: 10.1002/cncr.32003. Epub 2019 Feb 12. PMID 30748006
- [Background] Li C, Wu M, Wang J, Zhang S, Zhu L, Pan J, Zhang W. A population-based study on the risks of cervical lesion and human papillomavirus infection among women in Beijing, People's Republic of China. Cancer Epidemiol Biomarkers Prev. 2010 Oct;19(10):2655-64. doi: 10.1158/1055-9965.EPI-10-0212. Epub 2010 Aug 18. PMID 20719907
- [Background] Zhao FH, Lin MJ, Chen F, Hu SY, Zhang R, Belinson JL, Sellors JW, Franceschi S, Qiao YL, Castle PE; Cervical Cancer Screening Group in China. Performance of high-risk human papillomavirus DNA testing as a primary screen for cervical cancer: a pooled analysis of individual patient data from 17 population-based studies from China. Lancet Oncol. 2010 Dec;11(12):1160-71. doi: 10.1016/S1470-2045(10)70256-4. Epub 2010 Nov 11. PMID 21075054
- [Background] Li X, Xiang F, Dai J, Zhang T, Chen Z, Zhang M, Wu R, Kang X. Prevalence of cervicovaginal human papillomavirus infection and genotype distribution in Shanghai, China. Virol J. 2022 Sep 12;19(1):146. doi: 10.1186/s12985-022-01879-y. PMID 36096810